CLINICAL TRIAL: NCT05825092
Title: Effects of Early Testosterone Gel Administration on Physical Performance in the Critically Ill: a Randomised Double Blind Clinical Trial
Brief Title: Effects of Early Testosterone Gel Administration on Physical Performance in the Critically Ill
Acronym: TestICUs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC N 2018 BACHOUMAS
Record Dates: First submitted 2022-11-30; First posted 2023-04-24 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-04

CONDITIONS: Critical Illness
Keywords: Critical ill patient; Physical performance; Testosterone
MeSH Terms: conditions — Critical Illness | interventions — Testosterone; Muscle Strength

STUDY DESIGN:
Intervention Model Description: This is a prospective, phase II, multi-centre, double blind, randomised, controlled, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AndroGel® 1.62% (Active Comparator): AndroGel® will be applied daily to the upper arms/shoulders. AndroGel® will be administered within 24 hours after inclusion for a period of 28 days or until hospital discharge.
  For patients discharged from ICU before day 28, AndroGel® will be administered in hospital wards to complete the 28 days of treatment or until hospital discharge
  Interventions: Drug: Androgel Topical Product; Diagnostic Test: Physical performance; Diagnostic Test: Muscle strength; Diagnostic Test: Muscular mass; Diagnostic Test: Test: Functional status; Diagnostic Test: Oxygen muscular consumption
- Placebo gel will be the same gel without testosterone (Placebo Comparator): Placebo gel will be applied daily to the upper arms/shoulders. Placebo gel will be administered within 24 hours after inclusion for a period of 28 days or until hospital discharge. For patients discharged from ICU before day 28, Placebo gel will be administered in hospital wards to complete the 28 days of treatment or until hospital discharge
  Interventions: Drug: Placebo; Diagnostic Test: Physical performance; Diagnostic Test: Muscle strength; Diagnostic Test: Muscular mass; Diagnostic Test: Test: Functional status; Diagnostic Test: Oxygen muscular consumption

INTERVENTIONS:
Drug: Androgel Topical Product — AndroGel® will be applied daily to the upper arms/shoulders at 9:00 am. The daily dose will be 101.25 mg in men and 20.25 mg in women. AndroGel® will be administered within 24 hours after inclusion for a period of 28 days or until hospital discharge. For patients discharged from ICU before day 28, AndroGel® will be administered in hospital wards to complete the 28 days of treatment or until hospital discharge
  Other Names: Androgel 1.62% Transdermal Gel
  Arms: AndroGel® 1.62%
Drug: Placebo — Placebo gel will be applied daily to the upper arms/shoulders at 9:00 am. The daily dose will be 101.25 mg in men and 20.25 mg in women. Placebo gel will be administered within 24 hours after inclusion for a period of 28 days or until hospital discharge. For patients discharged from ICU before day 28, Placebo gel will be administered in hospital wards to complete the 28 days of
  Arms: Placebo gel will be the same gel without testosterone
Diagnostic Test: Physical performance — Physical performance at 3, 6 months and 1 year after ICU admission
  6 minute walk distance 3 months after ICU admission, at 6 months and at 1 year Percentage of patients with Short Physical Performance Battery < 10 at 3, 6 months and 1 year Physical component of SF 36 (Medical Outcomes Study 36 Item Short Form Health Survey) at 3, 6 months and 1 year
Diagnostic Test: Muscle strength — Muscle strength at ICU discharge at 3, 6 months and 1 year after ICU admission
  Handgrip: Kg and percent of the predicted force Medical Research Council testing (MRC)
Diagnostic Test: Muscular mass — Muscular mass at 3, 6 months and 1 year after ICU admission
  Mid-arm muscle circumference (MAMC)
Diagnostic Test: Test: Functional status — Functional status at 3, 6 months and 1 year after ICU admission
  • Composite score of 11 items of Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL)
Diagnostic Test: Oxygen muscular consumption — Oxygen muscular consumption at ICU discharge and at 3 months after ICU admission
  Ventilation free days at day 28 Length of stay in ICU Length of stay in hospital Mortality rate at day 28 Mortality rate at day 90 ICU mortality rate Hospital mortality rate

SUMMARY:
Critically ill patients experience major insults that lead to increased protein catabolism.

Hypermetabolism occurs early and rapidly during the first week of critical illness to provide amino acids for the production of energy via gluconeogenesis, and also for the synthesis of acute phase proteins and repair of tissue damage. During acute phase, neuroendocrine and inflammatory responses promote protein breakdown and amino acid release. Under stress conditions, protein synthesis cannot match the increased rate of muscle proteolysis because of a state of anabolism resistance, which limits uptake of amino acids into muscles.

Hypermetabolism results in a significant loss of lean body mass with an impact on weaning from the ventilator and muscle recovery. Functional disability can be long term sometimes with no full return to normal.

In critically ill patients, severe and persistent testosterone deficiency is very common and is observed early after Intensive Care Unit (ICU) admission. This acquired hypogonadism promotes the persistent loss of skeletal muscle protein and is related to poor outcome.

Administration of testosterone induces skeletal muscle fiber hypertrophy and decreases protein breakdown in healthy young men. It has been repeatedly shown that testosterone treatment enhances muscle mass and strength in hypogonadal men and women and can improve physical performance. Testosterone administration in burned patients reduces protein breakdown and increases protein synthesis efficiency. Oxandrolone, a synthetic testosterone analogue, reduces body mass and nitrogen loss and accelerates healing in burned patients. Trials in critically ill unburned patients failed to demonstrate any effect on clinical outcome but the studies were underpowered to detect a difference.

Transdermal gel testosterone is the preferred route of administration for achieving steady serum testosterone concentrations as compared to oral and intramuscular formulations.

Intramuscular injection induces strong fluctuations of testosterone plasma concentrations and can cause haematoma in patients with coagulation disorders, a common condition in ICUs. Several studies have raised the concern that testosterone administration could increase the risk of cardiovascular disease events. However, in a recent meta-analysis, no significant effects on cardiovascular risk were observed with either injected or transdermal testosterone supplementation in men, and the French National Agency for Medicines (ANSM) recently reported that drugs containing testosterone were not associated with an increased risk of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged over 18 years
* Negative pregnancy test (b-HCG) in female patient of childbearing potential
* Invasive mechanical ventilation expected to be required for more than 48 hours
* Written informed consent obtained from the patient or his/her legal representative
* Social security cover
* Contraception
* Female patient of childbearing potential (entering the study after a menstrual period and who has a negative pregnancy test), who agrees to use a highly effective method of contraception and an effective method of contraception by her male partner during treatment and for 7 months after the last treatment intake
* Male patient with a female partner of childbearing potential who agrees to use a highly effective method of contraception and an effective method of contraception by his female partner during treatment and for 4 months after the last treatment intake OR who agrees to use an effective method of contraception and a highly effective method of contraception by his female partner during the study and for 4 months after the last treatment intake

Exclusion Criteria:

* History of prostate cancer
* History of breast cancer
* Prostate cancer suspected or confirmed
* Breast cancer suspected or confirmed
* PSA (prostatic specific antigen) ≥ 4 ng/ml
* ICU length of stay > 120 h before enrollment
* Moribund
* Pre-existing illness with a life expectancy of <6 months
* Recent intracranial or spinal cord injury (< 1 month)
* Recent haemorrhagic or ischemic stroke (< 1 month)
* Neuromuscular disease
* Cardiac arrest in non-shockable rhythm
* Preexistent cognitive impairment or language barrier
* Inability to walk without assistance prior to acute ICU illness (use of a cane or walkers not excluded)
* Documented allergy to testosterone
* Age > 80 years
* Pregnancy
* Breast feeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
the 6-minute-walk distance test (6MWD) | 3 months after ICU admission
  Physical performance 3 months after ICU admission assessed by the 6-minute-walk distance test (6MWD) in metres. Absolute values will be compared to show a minimum absolute difference of 30 meters

SECONDARY OUTCOMES:
the 6-minute-walk | 6 months
  Percentage of patients with 6 MWD at 6 months > 60% the distance walked in an age-matched and sex-matched control population
the 6-minute-walk | 1 year after ICU admission
  Percentage of patients with 6 MWD at 1 year > 65% the distance walked in an age-matched and sex-matched control population
Functional status with Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) | at 3, 6 months and 1 year after ICU admission
  11 items of Activities of Daily Living (ADL) and Instrumental
  Activities of Daily Living (IADL):
Oxygen muscular consumption with NIRS test (Near Infrared Spectroscopy) | 48 hours after intensive care unit (ICU) admission and 3 months after ICU admission
  Low muscle oxidative capacity is associated with muscle dysfunction and exercise intolerance in COPD patients and may contribute to reduce physical activity and quality of life in these patients. Muscle maximal oxidative capacity can be evaluated by oxygen muscular consumption which will be measured by Near Infrared Spectroscopy (NIRS), during a series of short arterial occlusions in muscle quadriceps. Studies performed in healthy subjects showed a good agreement with high-resolution respirometry and phosphorus magnetic resonance spectroscopy (P-MRS) for assessing mitochondrial respiratory capacity. In COPD patients, NIRS technique was feasible and well tolerated.
Muscular mass with MAMC (Mid-arm muscle circumference): | at 3, 6 months and 1 year after ICU admission
  Mid-arm muscle circumference (MAMC) : MAMC (Mid-arm muscle circumference): MAMC is calculated using the following formula:
  MAMC = mid-arm circumference - (3.14 × triceps skinfold thickness). The mid-arm circumference is measured using a standard flexible measuring tape on the left upper arm, at the mid-point between the olecranon process of the shoulder and the acromion, with the subject in a seated position. The triceps skinfold thickness is measured using a calibrated skinfold caliper (range 0.00- 50.00 mm; minimum graduation 0.2 mm) (85).
the Short Physical Performance Battery (SPPB) | 3, 6 months and 1 year after ICU admission
  Percentage of patients with Short Physical Performance Battery < 10 at 3 months: The SPPB represents the sum of results from three component tests of functional relevance: standing balance, 4-meter gait speed (4MGS), and fiverepetition sit-to-stand motion (5STS). Each component is scored based on a subscale, and the three subscores are added to obtain a summary score. The SPPB is a high-level physical function outcome as it examines gait speed, balance control and sit-to-stand repetitions. It has been commonly used in COPD patients. In critical ill patients, the SPPB may be more appropriate as a measure in the post ICU setting in the acute hospital wards or post hospital discharge.
Physical component of Medical Outcomes Study 36 Item Short Form Health (SF36) | 3, 6 months and 1 year after ICU admission
  Physical component of SF 36 (Medical Outcomes Study 36 Item Short Form Health):
  The physical component of SF 36 is a commonly used and well validated instrument in critical ill patients. The SF 36 has demonstrated reliability, validity and responsiveness and is recommended in ICU populations.
Muscle strength by Handgrip test | 48 hours after ICU admission, at 3, 6 months and 1 year after ICU admission
  Kg and percent of the predicted force: Hand-grip strength (HGS) is a manual muscle test that enables measurement of force using a calibrated device. It is reliable, rapid and simple and can serve as a surrogate for global strength. Normative data are available. HGS has been commonly used in critical ill patients.
Muscle strength by Medical Research Council (MRC) score | at 3, 6 months and 1 year after ICU admission
  MRC has been routinely used in critical care research to screen for muscle weakness. It classifies muscle contraction on a 0-5 point ordinal scale. Six muscle groups will be assessed bilaterally.
Ventilation free days | at day 28
  Number of day without ventilation
Length of stay in the ICU | 48 hours after ICU admission
  Number of date between ICU admission and ICU discharge
Length of stay in hospital | at hospital discharge, an average of 1 month
  Number of date between ICU admission and hospital discharge
Mortality rate at day 28 | at day 28
  rate of patient included in the study and died at day 28
Mortality rate at day 90 | at day 90
  rate of patient included in the study and died at day 90
ICU mortality rate | 48 hours after ICU admission
  rate of patient included in the study and died at ICU discharge
Hospital mortality rate | at hospital discharge, an average of 1 month
  rate of patient included in the study and died at hospital discharge
Nombers of adverses events | from day 1 to day 28
  Safety of testosterone gel

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos BACHOUMAS, MD, Principal Investigator — Hospital, La Roche sur Yon; Bertrand SOUWEINE, MD, PhD, Study Director — University Hospital, Clermont-Ferrand
Locations (5):
- France (5):
  - Service de Medecine Intensive et Réanimation CHU de Bordeaux Hopital Pellegrin, Bordeaux
  - Service d'Anesthésie et Réanimation Centre Jean-Perrin, Clermont-Ferrand
  - Service de Médecine Intensive et Réanimation (MIR), CHU Clermont-Ferrand, Clermont-Ferrand
  - Service de Médecine Intensive et de Réanimation CHD La Roche sur Yon, La Roche-sur-Yon
  - Service de Médecine Intensive et Réanimation CHU Nantes, Hôtel Dieux, Nantes